CLINICAL TRIAL: NCT00627484
Title: Changes in Insulin Sensitivity After Weight Loss Induced by Diet or Bariatric Surgery
Brief Title: Changes in Insulin Sensitivity After Weight Loss
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Judith Korner, Associate Professor of Medicine, Columbia University
Other Study IDs: AAAB2401; R21DK081050 (NIH); DK072011 (Other Grant/Funding Number: NIDDK)
Record Dates: First submitted 2008-02-28; First posted 2008-03-03 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Obesity; Type 2 Diabetes Mellitus; Insulin Resistance
Keywords: Insulin resistance; Insulin sensitivity; bariatric surgery; diabetes; calorie restriction; body composition
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance; Diabetes Mellitus | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The researchers may want to retain your blood and/or tissue sample(s) so that additional research studies can be done now or in the future.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Group 1: GBP non-diabetic: Non-diabetic subjects scheduled to receive gastric bypass
  Interventions: Procedure: Gastric bypass
- Group 2: BND non-diabetic: Non-diabetic subjects scheduled to receive gastric banding
  Interventions: Procedure: Gastric banding
- Group 3: GBP diabetic: Diabetic subjects scheduled to receive gastric bypass
  Interventions: Procedure: Gastric bypass
- Group 4: VLCD diabetic: Diabetic subjects scheduled to receive very low calorie diet
  Interventions: Behavioral: Very low calorie diet
- Group 5: SG diabetic: Diabetic subjects scheduled to receive sleeve gastrectomy
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Gastric bypass — NOTE: the surgery is not paid for by the study
  Other Names: GBP
  Groups: Group 1: GBP non-diabetic; Group 3: GBP diabetic
Procedure: Gastric banding — NOTE: the surgery is not paid for by the study
  Other Names: BND
  Groups: Group 2: BND non-diabetic
Procedure: Sleeve gastrectomy — NOTE: the surgery is not paid for by the study
  Other Names: SG
  Groups: Group 5: SG diabetic
Behavioral: Very low calorie diet — Weight loss with calorie restricted liquid diet. Subject will be asked to stay in our in-patient research unit for 2-3 weeks and consume only those foods supplied by our bionutrition unit. Expected weight loss should be between 7-10% of body weight. Subjects will receive the diet at no cost and will be compensated for their time.
  Other Names: VLCD
  Groups: Group 4: VLCD diabetic

SUMMARY:
This study is designed to compare the changes in insulin sensitivity as well as gastrointestinal hormone levels in diabetic and non-diabetic obese individuals who are undergoing weight loss procedures. The main hypothesis of this study is that weight loss induced by gastric bypass will induce a greater improvement in insulin sensitivity compared with gastric banding or low calorie diet. Subjects will be studied before and after weight loss. Studies consist of intravenous glucose tolerance test, body composition analysis, meal test, and energy expenditure.

DETAILED DESCRIPTION:
Patients who are scheduled for gastric bypass (GBP), sleeve gastrectomy (SG), or simple caloric restriction with gastric banding (BND) or a very low calorie diet (VLCD) will be examined at baseline weight, and when 6-10% total body weight has been lost. We will measure insulin sensitivity with an intravenous glucose tolerance test, and fasting levels of hormones that regulate food intake and insulin sensitivity, such as ghrelin, peptide YY (PYY), glucagon-like peptide 1 (GLP1) and leptin. Fat mass and skeletal muscle mass will be measured by dual photon absorptiometry (DXA). We will also measure the hormonal and thermic response to food with a liquid test meal and energy expenditure by indirect calorimetry. This measures how many calories are burned at rest and the in response to food. Subjects with diabetes will continue to be studied with the same protocol on an annual basis out to 5 years in order to determine the rate of remission of diabetes and the durability of this effect as subjects tend to regain some body weight over time.

Subjects with diabetes will also be followed every three months for the first year after the initial weight loss for HbA1c and fasting glucose levels. The results of this study may lead to new understanding about changes in insulin sensitivity, body composition and hormonal profile, as well as changes in energy expenditure with weight loss after bariatric surgery or with simple caloric restriction. With this greater understanding, new treatments for obesity and diabetes, that do not require surgery, may be developed.

ELIGIBILITY:
Inclusion criteria:

* Non-diabetic obese (BMI > 30) adult men and women between the ages of 18 and 75 scheduled to undergo

  * gastric bypass (GBP)
  * gastric banding (BND)
* Type 2 diabetes (HbA1c 6-12%) adult men and women between the ages of 18 and 75 scheduled to undergo gastric bypass.
* Type 2 diabetes (HbA1c 6-12%) adult men and women between the ages of 18 and 65 for weight reduction with a very low caloric diet (VLCD).
* Type 2 diabetes mellitus scheduled to undergo sleeve gastrectomy (SG).

Exclusion criteria:

* Pregnancy.
* Age > 75 for surgery groups; Age > 65 for VLCD group.
* Treatment with glucocorticoids, anti-depressants, anti-psychotics, neuroleptics, weight loss medications, experimental medication.
* Greater than a 5% change in total body weight in the 90 days prior to the study.
* History of untreated gallstones; hepatic or renal insufficiency, abnormal thyroid stimulating hormone (TSH).
* Use of thiazolidinedione therapy.
* HbA1c > 12%.
* Use of dipeptidyl peptidase IV (DPP-IV) inhibitor or glucagon-like peptide 1 receptor (GLP-1R) agonist for greater than 12 months within 3 months of the study.
* Fasting triglycerides > 400.
* Significant cardiovascular, neurologic, renal, gastrointestinal, or hematologic disease.
* Inability to comply with or understand the study protocol as ascertained by the PI.
* We will not exclude individuals with body weight > 145 kg, but we do recognize that such individuals are above the table weight limitations of the dual-energy x-ray absorptiometry (DEXA) scan and body composition data will be unavailable for those individuals.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited by physician referral and from outpatient obesity, bariatric surgical clinics and endocrinology clinics at Columbia University Medical Center as well as from the Medical Center Community and metropolitan area via IRB-approved flyers and internet postings. Subjects will also be recruited from the following website: www.craigslist.com using the same posting format of the IRB-approved flyers.
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2005-03-01 (Actual); Primary Completion 2018-06-17 (Actual); Study Completion 2018-06-17 (Actual)

PRIMARY OUTCOMES:
Change in Insulin Sensitivity | 2-8 weeks
  Measured by frequently sampled intravenous glucose tolerance test (FSIVGTT)

SECONDARY OUTCOMES:
Change in Body Composition | 2-8 weeks
  Measured by dual energy x-ray absorptiometry (DXA)
Change in Resting Energy Expenditure | Up to 4 hrs post-meal
  Measured by indirect calorimetry using a Hood Calorimeter

CONTACTS AND LOCATIONS:
Overall Officials: Judith Korner, MD,PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jackness C, Karmally W, Febres G, Conwell IM, Ahmed L, Bessler M, McMahon DJ, Korner J. Very low-calorie diet mimics the early beneficial effect of Roux-en-Y gastric bypass on insulin sensitivity and beta-cell Function in type 2 diabetic patients. Diabetes. 2013 Sep;62(9):3027-32. doi: 10.2337/db12-1762. Epub 2013 Apr 22. PMID 23610060